CLINICAL TRIAL: NCT03658577
Title: Association of Beta-Blocker Therapy at Discharge With Clinical Outcomes in Patients With Actue Coronary Syndrome Undergoing Percutaneous Coronary Intervention
Brief Title: Association of Beta-Blocker Therapy at Discharge With Clinical Outcomes in Patients With Actue Coronary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: COE20180821
Record Dates: First submitted 2018-08-20; First posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Actue Coronary Syndrome
Keywords: Actue Coronary Syndrome; Beta-Blocker; Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Limited data are available on the efficacy of beta-blocker therapy for secondary prevention in Actue Coronary Syndrome(ACS) patients. This study sought to investigate the association of beta-blocker therapy at discharge with clinical outcomes in patients with ACS after percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
The American College of Cardiology (ACC)/American Heart Association (AHA) guidelines recommend beta-blockers for secondary prevention in patients with ACS without regard to reperfusion therapy. However, evidence supporting this recommendation originated from studies conducted before the introduction of reperfusion therapy or studies in patients treated with fibrinolysis. In the present era of PCI, there are no prospective randomized studies looking at the effects of long-term beta-blocker therapy on clinical outcomes in ACS patients. Moreover, results from registry data and post-hoc analysis on beta-blocker therapy in patients undergoing PCI are inconsistent.

In particular, the beneficial effect of long-term beta-blocker therapy has not been well established in patients with relatively low risk, such as preserved left ventricular systolic function or single-vessel disease. Therefore, we investigated the association of beta-blocker therapy at discharge with clinical outcomes in ACS patients after PCI.

ELIGIBILITY:
Inclusion Criteria:

1. consecutive patients 18 years of age or older;
2. patients diagnosed as ACS(including STEMI、NSTEMI and UA) by doctor at discharge;
3. patients undergoing primary PCI.

Exclusion Criteria:

missing beta-blocker information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was selected from ten major cardiac centres in ShenZhen,CHINA.
Sampling Method: Probability Sample
Enrollment: 582 (Estimated)
Dates: Start 2018-03-02 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
all-cause death | 3 years
  The primary outcome was all-cause death during follow up.

SECONDARY OUTCOMES:
MACE | 3 year
  Secondary outcomes included major adverse cardiac events (MACE), a composite of cardiac death, myocardial infarction, stroke, any revascularization during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: ShaoHong P Dong, PhD, Principal Investigator — professor, Chief of cardiovascular department
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided